CLINICAL TRIAL: NCT03941769
Title: A Phase I/II Study of Recombinant Human Interleukin-7 to Promote T-Cell Recovery After Haploidentical and Cord Blood Stem Cell Transplantation
Brief Title: 2018-0674 - IL-7 for T-Cell Recovery Post Haplo and CB Transplant - Phase I/II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0674; NCI-2019-02124 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0674 (Other: M D Anderson Cancer Center); R01CA061508 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Cord Blood Transplant Recipient; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (recombinant interleukin-7) (Experimental): Within 60-180 days after CBT, patients receive recombinant interleukin-7 IM or SC once per week for 3 weeks.
  Interventions: Biological: Recombinant Interleukin-7

INTERVENTIONS:
Biological: Recombinant Interleukin-7 — Given IM or SC
  Other Names: CYT 99 007; CYT-107; IL-7; Lymphopoietin-1; Recombinant Human Interleukin-7

SUMMARY:
This phase I/II trial studies side effects and best dose of recombinant interleukin-7 in promoting immune cell recovery in patients with acute myeloid leukemia, myelodysplastic syndrome, chronic myeloid leukemia, or myeloproliferative disease after a haploidentical or cord blood stem cell transplant. A haploidentical transplant is a transplant that uses stem cells from a donor that is partially (at least 50%) matched to the patient. Umbilical cord blood is a source of blood-forming cells that can be used for transplant, also known as a graft. However, there is a small number of blood-forming cells available in the transplant, which may delay the "take" of the graft in the recipient. Recombinant interleukin-7 may affect the "take" of the graft and the recovery of certain blood cells related to the immune system (called T-cells, natural killer cells, and B cells) in patients who have had a haploidentical or cord blood stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and establish the optimal biologic dose of glycosylated recombinant human interleukin-7 (CYT107).

SECONDARY OBJECTIVES:

I. To determine the rate of cytomegalovirus (CMV), Epstein-Barr virus (EBV) and BK viral infections in umbilical cord blood stem cell transplantation (CBT) and haploidentical stem cell transplantation (haplo-SCT) patients who receive three doses of interleukin-7 (IL-7) following engraftment.

II. To calculate the overall survival (OS), progression-free survival (PFS), and cumulative incidence of graft versus host disease (GVHD) and cumulative incidence of relapse.

III. To evaluate the effects of CYT107 on the recovery of T, natural killer (NK) and B cell populations and their functions in vitro; these data will be used to identify the optimal dose to move to a phase II trial.

OUTLINE: This is a dose-escalation study.

Within 60-180 days after CBT, patients receive recombinant interleukin-7 intramuscularly (IM) or subcutaneously (SC) once per week for 3 weeks.

After completion of study treatment, patients are followed for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* English and non-English speaking patients are eligible.
* Patient post a cord blood transplant (CBT) or haplo-SCT, with matched unrelated donors (MUDs), both peripheral blood (PB) and marrow sources with documented absolute neutrophil engraftment
* Patients with documented engraftment but require granulocyte-colony stimulating factor (G-CSF) to treat myelosuppression induced by drugs used to treat or prevent infection are eligible
* Karnofsky performance status (KPS) > 60%
* Absence of dyspnea or hypoxia (< 90% of saturation by pulse oximetry on room air)
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Prothrombin time (PT)/partial prothrombin time (PTT) < 1.5 x ULN
* Calculated creatinine clearance > 60 mL/min/1.73 m^2
* Diagnosis of acute myeloid leukemia; myelodysplastic syndrome; chronic myeloid leukemia; myelofibrosis or myeloproliferative disease

Exclusion Criteria:

* Pregnant or nursing
* History of lymphoid malignancy (including Hodgkin disease, non-Hodgkin lymphoma, acute lymphoblastic leukemia and chronic lymphocytic leukemia) or acute biphenotypic leukemia
* Patients with acute GVHD > grade 2 at any time during the post-transplant course
* Ongoing immunosuppressive therapy for the treatment of GVHD. Patients receiving GVHD prophylaxis will be allowed on this study
* History of Epstein-Barr virus (EBV) associated lymphoproliferation
* Active uncontrolled viral, bacterial or fungal infection
* History of autoimmune disease
* Receiving systemic corticosteroid therapy, budesonide is allowed
* Uncontrolled hypertension
* Corrected QT (QTc) prolongation (QTc > 470 ms) or prior history of significant arrhythmia or electrocardiogram (ECG) abnormalities
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Patients with cognitive impairments and/or any past or current psychiatric illness that, in the opinion of the investigator, would interfere with adherence to study requirements or the ability and willingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gheath Al-Atrash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Supportive Care (Recombinant Interleukin-7)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Recombinant Interleukin-7)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Participants that had grade 3 or 4 graft versus host disease (GVHD), secondary graft failure, disease relapse, development of post-transplant lymphoproliferative disorder, development of progressive multifocal leukoencephalopathy or grade 3-4 organ failure attributable to recombinant human interleukin-7 (CYT107) and death.
Time Frame: Up to 42 days after first injection
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Recombinant Interleukin-7)
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Overall Survival
Description: Number of participant that survived after 3 years.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Recombinant Interleukin-7)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 42 days from the last injection of CYT107, up to 3 years
Arm/Group | Supportive Care (Recombinant Interleukin-7)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Recombinant Interleukin-7) (N=1)
White blood cell decreased (Investigations) | 1
Increased ALT (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
ANC Decreased (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03941769/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT03941769/ICF_001.pdf